CLINICAL TRIAL: NCT05701852
Title: Motivational Behavioral and Functional MRI Impairment in Patients With Chronic Neuropathic Pain
Acronym: MOTION
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: HBD_2022_6
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases : patients with chronic pain
  Interventions: Other: reward learning task
- controls
  Interventions: Other: reward learning task

INTERVENTIONS:
Other: reward learning task — during usual follow-up patients will complete a remard learning task questionnaire. This questionnaire cannot be assimilated to a clinical intervention.

SUMMARY:
The main hypothesis of this study is that the alteration of the reward circuitry underlying the motivational deficit in chronic pain patients compared to healthy subjects results in a decrease in the capacity for reward learning. The fMRI studies have shown that this type of learning depends on the dopaminergic system innervating key regions of the reward system.

ELIGIBILITY:
Inclusion Criteria:

* For cases: patients managed in the neurosurgery department or at CETD for chronic neuropathic pain, of central or peripheral origin.
* For controls: matched to a case on age (±5 years) and sex

Exclusion Criteria:

* Neurodegenerative or inflammatory neurological pathology
* Clinical depressive syndrome
* High doses of opioid treatment (greater than 100 mg/day of morphine equivalent)
* Impaired judgment or inability to receive information that does not allow the performance of behavioral tasks
* Absolute contraindication to MRI (e.g. pacemaker, implantable pacemaker, metallic intra-orbital foreign body)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to patients followed at the pain treatment center or in neurosurgery for chronic neuropathic pain, of peripheral or central origin.
  Controls will be recruited among the patients' companions and the staff of the Adolphe de Rothschild Foundation Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
To compare reward learning ability in patients with chronic neuropathic pain compared with an age (±5 years) and gender-matched control population | Day 0
  the reward learning ability will be assessed using a specific task. The result of the task questionnaire is a numeric score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No